CLINICAL TRIAL: NCT04963413
Title: RENEW: Pilot Study of Feasibility of CMV RNA-Pulsed Dendritic Cells Vaccines for the Treatment of Newly Diagnosed Glioblastoma Patients.
Brief Title: RENEW: Feasibility of CMV RNA-Pulsed Dendritic Cells Vaccines for the Treatment of Newly Diagnosed Glioblastoma Patients.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by mutual agreement by sponsor and institution.
Sponsor: University of Florida (Other)
Collaborators: Immunomic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202002778; OCR39689 (Other: OnCore)
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
Keywords: Immunotherapy; Vaccine Therapy; Immune system; Dendritic Cell; High grade brain tumor
MeSH Terms: conditions — Glioblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous DCs derived from PBMC loaded with RNA (Experimental): Autologous DCs derived from PBMC loaded with RNA encoding the human CMV matrix protein pp65-flLAMP plus GM-CSF
  Interventions: Biological: Autologous DCs derived from PBMC loaded with RNA encoding the human CMV matrix protein pp65-flLAMP plus GM-CSF

INTERVENTIONS:
Biological: Autologous DCs derived from PBMC loaded with RNA encoding the human CMV matrix protein pp65-flLAMP plus GM-CSF — Autologous DCs derived from PBMC loaded with RNA encoding the human CMV matrix protein pp65-flLAMP plus GM-CSF

SUMMARY:
In prior trials of CMV RNA-pulsed dendritic cell vaccines, there has been a narrow window between surgery and initiation of chemoradiation to enroll patients and perform leukapheresis (to obtain cells needed to generate investigational vaccine). Patients who had started chemoradiation were not eligible to participate.

In this study, the investigators propose to conduct a pilot study to evaluate the ability to generate pp65 full-length LAMP RNA-pulsed DCs in patients who have completed standard external beam radiation and concomitant temozolomide who are receiving adjuvant temozolomide chemotherapy at the time of enrollment.

DETAILED DESCRIPTION:
This pilot study will enroll adult patients with newly diagnosed WHO Grade IV glioma (GBM) who have completed standard of care chemoradiation and are receiving adjuvant temozolomide chemotherapy. Patients will undergo leukapheresis and resume their adjuvant chemotherapy cycles following their treatment plan for 1 to 2 cycles while CMV pp65 RNA-pulsed DCs are generated.

After QA/QC release, study Vaccine #1 will be given at day 22-24 of the TMZ cycle. All patients will receive Td booster (5 Lf) with Vaccine #1 regardless of booster history. Vaccine #2 and #3 will occur at 2-week intervals.

The following TMZ cycle will start about 2 weeks after Vaccine #3. Patients may complete up to 6 to 12 adjuvant cycles every 5 weeks with pp65 full-length RNA-pulsed DCs administered at day 22-24 of each cycle until all available vaccines are exhausted with a maximum of 10 study vaccines or until disease progression (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed diagnosis of de novo Glioblastoma (WHO Grade IV glioma) by histopathology or molecular studies. (Secondary GBM not eligible).
* The tumor must have a supratentorial component.
* Patient have completed standard external beam radiation with concomitant temozolomide.

(Minimum dose for concomitant radiotherapy is 40 Gy)

* Patient must be receiving adjuvant therapy with Temozolomide at time of enrollment.
* Karnofsky Performance Status (KPS) ≥ 70.
* Signed informed consent. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the legally authorized representative.
* For females of childbearing potential, negative serum pregnancy test at enrollment.
* Women of childbearing potential (WOCBP) must be willing to use acceptable contraceptive method to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.

Refer to Appendix B for definition of WOCBP and guidance on acceptable contraceptive methods.

-Males with female partners of childbearing potential must agree to practice adequate contraceptive methods throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

Refer to Appendix B for guidance on acceptable contraceptive methods.

* For patients receiving steroids, daily dose must be < 4 mg.
* Adequate Bone marrow and organ function as defined below:

  1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3.
  2. Platelet count ≥ 100,000 cells/mm3.
  3. Hemoglobin ≥ 9 g/dl. (The use of transfusion or other intervention to achieve Hgb ≥ 9 g/dl is acceptable.)
  4. BUN ≤ 25 mg/dl
  5. Creatinine ≤ 1.7 mg/dl
  6. Bilirubin ≤ 2.0 mg/dl
  7. ALT ≤ 5 times institutional upper limits of normal for age
  8. AST ≤ 5 times institutional upper limits of normal for age

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years.
* Metastases detected below the tentorium or beyond the cranial vault and leptomeningeal involvement.
* Recurrent disease
* Multifocal gliomas defined as distinct tumors that do not have overlapping T2/FLAIR signal.
* HIV, Hepatitis B, or Hepatitis C seropositive.
* Known active infection (requiring treatment by antiviral or antibiotic) at time of enrollment
* Immunosuppressive disease.
* Severe, active co-morbidity, defined as follows:

  1. Unstable angina and/or congestive heart failure requiring hospitalization.
  2. Transmural myocardial infarction within the last 6 months.
  3. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at initiation of XRT/TMZ.
  4. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  5. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  6. Patients with autoimmune disease requiring medical management with systemic immunosuppressants.
  7. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy.
* Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant.
* Women of childbearing potential and men who are sexually active and are unwilling or unable to use an acceptable method of contraception for the entire study; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Prior allergic reaction to TMZ, GM-CSF, or Td.
* Patients who have received an investigational agent within 28 days prior to study entry.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Ability to generate CMV pp65 RNA-pulsed DCs in patients receiving adjuvant temozolomide chemotherapy after radiotherapy. | Leukapheresis to investigational product release date or up to 6 weeks
  Proportion of patients who are able to generate at least 3 CMV pp65 RNA-pulsed DCs vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Shands Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No